CLINICAL TRIAL: NCT00337571
Title: A Multicenter Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study With Three Fixed Doses of Aripiprazole in the Treatment of Children and Adolescents With Autistic Disorder (AD)
Brief Title: Study of Aripiprazole in the Treatment of Children and Adolescents With Autistic Disorder (AD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CN138-179
Record Dates: First submitted 2006-06-13; First posted 2006-06-16 (Estimated); Results first posted 2009-07-23 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2009-11

CONDITIONS: Behavioral Symptoms; Autistic Disorder
Keywords: Serious behavioral problems in children and adolescents with AD
MeSH Terms: conditions — Behavioral Symptoms; Autistic Disorder | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A1 (Experimental): 5 mg
  Interventions: Drug: Aripiprazole
- A2 (Experimental): 10 mg
  Interventions: Drug: Aripiprazole
- A3 (Experimental): 15 mg
  Interventions: Drug: Aripiprazole
- B1 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — Tablets, Oral, once daily, 8 weeks
  Other Names: Abilify
  Arms: A1; A2; A3
Drug: Placebo — Tablets, Oral, once daily, 8 weeks
  Arms: B1

SUMMARY:
This study will compare the effectiveness (how well the drug works) of aripiprazole with placebo (fixed dose) in reducing serious behavioral problems in children and adolescents with a diagnosis of autistic disorder (AD).

ELIGIBILITY:
Inclusion Criteria:

* Meets current Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) diagnostic criteria for AD and demonstrates serious behavioral problems; diagnosis confirmed by Autism, Diagnostic Interview-Revised (ADI-R).
* CGI score > = 4 AND an ABC Irritability/Agitation subscale score > = 18 at screening and baseline (randomization)
* Mental age of at least 18 months
* Male or female 6 to 17 years of age inclusive, at the time of randomization

Exclusion Criteria:

* Patients considered treatment resistant to neuroleptic medication based on lack of therapeutic response to 2 different neuroleptics after treatment of at least 3 weeks each
* Patients previously treated and not responding to aripiprazole treatment
* The patient is currently diagnosed with another disorder on the autism spectrum, including PDD-NOS, Asperger's Disorder, Rett's Disorder, Fragile-X Syndrome or Childhood Disintegrative Disorder
* Current diagnosis of bipolar disorder, psychosis, schizophrenia, or major depression
* A seizure in the past year
* History of severe head trauma or stroke
* Non-pharmacologic therapy (e.g., psychotherapy, behavior modification) should be stable prior to screening and consistent throughout the study

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 218 (Actual)
Dates: Start 2006-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (31):
- United States (31):
  - University Of Alabama At Birmingham, Birmingham, Alabama
  - Harmonex Neuroscience, Dothan, Alabama
  - Southwest Autism Research And Resource Center, Phoenix, Arizona
  - Clinical Innovations, Inc., Huntington Beach, California
  - University Of California-Davis Medical Center, Sacramento, California
  - Stanford University School Of Medicine, Stanford, California
  - The Children'S Hospital, Aurora, Colorado
  - Marsella, Gregory, Boca Raton, Florida
  - University Of Florida, Gainesville, Florida
  - University Of South Florida, Tampa, Florida
  - Institute For Behavioral Medicine, Smyrna, Georgia
  - University Of Illinois At Chicago, Chicago, Illinois
  - Cambridge Health Alliance, Medford, Massachusetts
  - Ladders Clinic, Wellsley, Massachusetts
  - Children'S Hospital Of Michigan, Detroit, Michigan
  - Regions Hospital, Saint Paul, Minnesota
  - Children'S Mercy Hospital, Kansas City, Missouri
  - Munroe-Meyer Institute, Omaha, Nebraska
  - North Shore - Long Island Jewish Health System, Bethpage, New York
  - Seaver And New York Autism Center Of Excellence, New York, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Mission Hospitals, Asheville, North Carolina
  - Duke Child And Family Study Center, Durham, North Carolina
  - The Nisonger Center, Columbus, Ohio
  - Cutting Edge Research, Oklahoma City, Oklahoma
  - Western Psychiatric Institute And Clinic, Pittsburgh, Pennsylvania
  - Dallas Pediatric Neurology Associates, Dallas, Texas
  - Bayou City Research, Ltd., Houston, Texas
  - Children'S National Medical Center, Fairfax, Virginia
  - Pacific Institute Of Medical Sciences, Bothell, Washington
  - Children'S Hospital Of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Marcus RN, Owen R, Kamen L, Manos G, McQuade RD, Carson WH, Aman MG. A placebo-controlled, fixed-dose study of aripiprazole in children and adolescents with irritability associated with autistic disorder. J Am Acad Child Adolesc Psychiatry. 2009 Nov;48(11):1110-1119. doi: 10.1097/CHI.0b013e3181b76658. PMID 19797985
- [Derived] Mankoski R, Stockton G, Manos G, Marler S, McQuade R, Forbes RA, Marcus R. Aripiprazole treatment of irritability associated with autistic disorder and the relationship between prior antipsychotic exposure, adverse events, and weight change. J Child Adolesc Psychopharmacol. 2013 Oct;23(8):572-6. doi: 10.1089/cap.2012.0075. PMID 24138011
- [Derived] Robb AS, Andersson C, Bellocchio EE, Manos G, Rojas-Fernandez C, Mathew S, Marcus R, Owen R, Mankoski R. Safety and tolerability of aripiprazole in the treatment of irritability associated with autistic disorder in pediatric subjects (6-17 years old):results from a pooled analysis of 2 studies. Prim Care Companion CNS Disord. 2011;13(1):PCC.10m01008. doi: 10.4088/PCC.10m01008gry. PMID 21731831

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Aripiprazole 5 mg | Aripiprazole 10 mg | Aripiprazole 15 mg
Started | 52 | 53 | 59 | 54
Completed | 38 | 44 | 49 | 47
Not Completed | 14 | 9 | 10 | 7
Not completed — Lack of Efficacy | 3 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 5 | 8 | 4
Not completed — Withdrawal by Subject | 2 | 2 | 1 | 0
Not completed — Lost to Follow-up | 3 | 1 | 0 | 1
Not completed — Poor/noncompliance | 1 | 1 | 1 | 1
Not completed — No longer met study criteria | 1 | 0 | 0 | 0
Not completed — High Potassium level | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Aripiprazole 5 mg | Aripiprazole 10 mg | Aripiprazole 15 mg | Total
Number analyzed (Participants) | 52 | 53 | 59 | 54 | 218
Age, Customized [Number; unit: participants]
  6 to 12 years | 35 | 44 | 45 | 42 | 166
  13 to 17 years | 17 | 9 | 14 | 12 | 52
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 9 | 4 | 23
  Male | 48 | 47 | 50 | 50 | 195
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 3 | 1 | 2 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 13 | 13 | 15 | 9 | 50
  White | 35 | 37 | 41 | 42 | 155
  Other | 1 | 2 | 1 | 2 | 6
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic/Latino | 8 | 5 | 7 | 5 | 25
  Not Hispanic/Latino | 44 | 48 | 52 | 49 | 193
Weight Group [Number; unit: Participants]
  <40 kilograms | 24 | 35 | 33 | 34 | 126
  ≥40 kilograms | 28 | 18 | 26 | 20 | 92
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 20.49 (4.777) | 19.91 (6.124) | 21.06 (6.649) | 20.14 (6.033) | 20.41 (5.933)
Height [Mean (Standard Deviation); unit: centimeters] | 144.9 (18.82) | 136.5 (14.66) | 142.3 (17.87) | 139.3 (17.24) | 140.8 (17.38)
Weight [Mean (Standard Deviation); unit: kilograms] | 45.6 (20.01) | 38.9 (18.26) | 44.8 (22.38) | 42.2 (22.99) | 42.9 (21.07)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change (Week 8 - Baseline) in the Autistic Behavior Checklist (ABC) Irritability Subscale Score
Description: The ABC is a 58-item informant-based assessment of problem behaviors in children/adolescents with mental retardation. Items are rated on a 4-point scale (0=no problem, 3=severe problem), and resolve into 5 domain subscales. A decrease in score indicates improvement.
Time Frame: Week 8
Population: Efficacy population=all randomized participants minus 3 patients in the placebo group (1 lost to follow-up, 1 withdrew consent, 1 no longer met study criteria), 1 participant in the 5-mg group who withdrew consent, and 1 participant in the 15-mg group who had elevated potassium levels. Data set is LOCF.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole 5 mg | Aripiprazole 10 mg | Aripiprazole 15 mg
Number analyzed (Participants) | 49 | 52 | 59 | 53
units on a scale | -8.4 (1.39) | -12.4 (1.36) | -13.2 (1.25) | -14.4 (1.31)

2. Secondary Outcome: Mean Clinical Global Impressions Improvement Scale (CGI-I) Score
Description: The CGI scale is a clinician-rated global assessment of a patient's improvement over time. Baseline assessment rated a patient's condition on a 7-point scale (1=no symptoms, 7=very severe symptoms). Subsequent assessed improvement relative to baseline symptoms on a 7-point CGI-I item scale (1=very much improved, 7=very much worse).
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole 5 mg | Aripiprazole 10 mg | Aripiprazole 15 mg
Number analyzed (Participants) | 49 | 52 | 59 | 53
units on a scale | 3.3 (0.18) | 2.6 (0.17) | 2.5 (0.16) | 2.5 (0.17)

3. Secondary Outcome: Number of Participants With Response at Week 8
Description: Response defined as a ≥ 25% reduction from baseline to endpoint in the ABC Irritability Subscale score and a CGI-I score of 1 or 2 at endpoint.
Time Frame: Week 8
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Placebo | Aripiprazole 5 mg | Aripiprazole 10 mg | Aripiprazole 15 mg
Number analyzed (Participants) | 49 | 52 | 59 | 53
Participants | 17 | 29 | 29 | 28

4. Secondary Outcome: Mean Change (Week 8 - Baseline) in the Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS; Compulsion Scale Only)
Description: CY-BOCS=10-item assessment of obsessive-compulsive symptoms in patients <18 years. 5 items pertaining to compulsions rate symptoms (time spent, interference with functioning, distress, resistance, control) on a 5-point scale (0=no symptoms/minimum severity, 4=extreme symptoms/maximum severity). A decreased in value indicates improvement.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole 5 mg | Aripiprazole 10 mg | Aripiprazole 15 mg
Number analyzed (Participants) | 44 | 46 | 54 | 48
units on a scale | -1.7 (0.50) | -2.6 (0.50) | -2.4 (0.44) | -3.2 (0.47)

5. Secondary Outcome: Mean Change (Week 8 - Baseline) in the Other ABC Subscale Scores
Description: Mean change (Week 8 - baseline) in the other ABC subscale scores (lethargy/social withdrawal; stereotypic behavior; hyperactivity/ noncompliance; inappropriate speech). A decrease in value indicates improvement.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole 5 mg | Aripiprazole 10 mg | Aripiprazole 15 mg
Number analyzed (Participants) | 49 | 52 | 59 | 53
units on a scale
  ABC Hyperactivity Subscale Score | -7.7 (1.67) | -14.0 (1.64) | -13.3 (1.50) | -16.3 (1.59)
  ABC Stereotypy Subscale Score | -1.8 (0.69) | -4.5 (0.68) | -4.2 (0.63) | -4.5 (0.66)
  ABC Inappropriate Speech Subscale Score | -1.1 (0.46) | -2.0 (0.45) | -1.8 (0.41) | -2.3 (0.43)
  ABC Social Withdrawal Subscale Score | -5.2 (1.16) | -5.8 (1.15) | -4.9 (1.06) | -7.9 (1.11)

6. Secondary Outcome: Mean Change (Week 8 - Baseline) in CGI-Severity (CGI-S)
Description: A CGI-S assessment (a 7-point scale to evaluate the severity of symptoms) was performed at baseline (1=no symptoms; 7=very severe symptoms). The patient's improvement relative to the symptoms at baseline on were assessed on a 7-point CGI-I (1=very much improved; 7=very much worse). A decrease in value indicates improvement.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Aripiprazole 5 mg | Aripiprazole 10 mg | Aripiprazole 15 mg
Number analyzed (Participants) | 41 | 44 | 52 | 44
units on a scale | -0.6 (0.16) | -0.9 (0.15) | -1.0 (0.13) | -1.1 (0.15)

7. Secondary Outcome: Summary of Safety
Description: Deaths, Adverse Events (AEs), Serious AEs (SAEs), Treatment-Emergent AEs and AEs leading to discontinuation
Time Frame: continuously throughout the study
Population: Safety population=all randomized participants minus 1 patients in the placebo group (no longer met study criteria), and 1 participant in the 5-mg group who withdrew consent.
Measure: Number; unit: participants
Arm/Group | Placebo | Aripiprazole 5 mg | Aripiprazole 10 mg | Aripiprazole 15 mg
Number analyzed (Participants) | 51 | 52 | 59 | 54
participants
  Deaths | 0 | 0 | 0 | 0
  Treatment-emergent SAEs | 0 | 1 | 1 | 0
  AEs leading to discontinuation of study medication | 4 | 5 | 8 | 4
  Treatment-emergent AEs overall | 37 | 46 | 53 | 46
  Treatment-emergent AEs related to study medication | 22 | 37 | 50 | 39
  Treatment-emergent extrapyramidal symptom AEs | 6 | 12 | 13 | 12

8. Secondary Outcome: Change From Baseline in Body Weight
Description: Adjusted mean change (Week 8 - baseline) in body weight
Time Frame: Week 8
Population: Safety population=all randomized participants minus 3 patients in the placebo group (1 no longer met study criteria, 2 did not have measurement at baseline and Week 8), and 1 participant in the 5-mg group who withdrew consent. Data set is LOCF.
Measure: Mean (Standard Error); unit: kilograms
Arm/Group | Placebo | Aripiprazole 5 mg | Aripiprazole 10 mg | Aripiprazole 15 mg
Number analyzed (Participants) | 49 | 52 | 59 | 53
kilograms | 0.3 (0.32) | 1.3 (0.31) | 1.3 (0.29) | 1.5 (0.30)

ADVERSE EVENTS:
Arm/Group | Aripiprazole 10 mg | Aripiprazole 15 mg | Aripiprazole 5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/59 | 0/54 | 1/52 | 0/51
Other Adverse Events (participants affected / at risk) | 51/59 | 42/54 | 37/52 | 31/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole 10 mg (N=59) | Aripiprazole 15 mg (N=54) | Aripiprazole 5 mg (N=52) | Placebo (N=51)
AGGRESSION (Psychiatric disorders) | 1 | 0 | 0 | 0
PRESYNCOPE (Nervous system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole 10 mg (N=59) | Aripiprazole 15 mg (N=54) | Aripiprazole 5 mg (N=52) | Placebo (N=51)
WEIGHT INCREASED (Investigations) | 1 | 2 | 4 | 1
INSOMNIA (Psychiatric disorders) | 5 | 2 | 1 | 6
AGGRESSION (Psychiatric disorders) | 2 | 0 | 2 | 3
SEASONAL ALLERGY (Immune system disorders) | 0 | 1 | 0 | 4
TREMOR (Nervous system disorders) | 7 | 6 | 4 | 0
DROOLING (Nervous system disorders) | 8 | 5 | 2 | 0
HEADACHE (Nervous system disorders) | 5 | 5 | 3 | 2
LETHARGY (Nervous system disorders) | 3 | 3 | 4 | 0
SEDATION (Nervous system disorders) | 17 | 13 | 9 | 3
AKATHISIA (Nervous system disorders) | 2 | 0 | 1 | 3
SOMNOLENCE (Nervous system disorders) | 5 | 5 | 4 | 2
HYPERSOMNIA (Nervous system disorders) | 0 | 2 | 3 | 0
EXTRAPYRAMIDAL DISORDER (Nervous system disorders) | 4 | 6 | 2 | 0
PSYCHOMOTOR HYPERACTIVITY (Nervous system disorders) | 0 | 0 | 3 | 2
NAUSEA (Gastrointestinal disorders) | 3 | 4 | 1 | 1
VOMITING (Gastrointestinal disorders) | 12 | 5 | 5 | 4
DIARRHOEA (Gastrointestinal disorders) | 5 | 5 | 2 | 4
CONSTIPATION (Gastrointestinal disorders) | 6 | 3 | 2 | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 4 | 2 | 1
SALIVARY HYPERSECRETION (Gastrointestinal disorders) | 4 | 6 | 1 | 1
NASOPHARYNGITIS (Infections and infestations) | 5 | 5 | 6 | 2
GASTROENTERITIS VIRAL (Infections and infestations) | 3 | 1 | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 3 | 2 | 0
ENURESIS (Renal and urinary disorders) | 1 | 3 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 5 | 3 | 5 | 1
INCREASED APPETITE (Metabolism and nutrition disorders) | 3 | 7 | 10 | 2
RASH (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 8 | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 2 | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 1
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3
THIRST (General disorders) | 1 | 1 | 3 | 1
FATIGUE (General disorders) | 13 | 10 | 2 | 0
PYREXIA (General disorders) | 7 | 5 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.